CLINICAL TRIAL: NCT05776511
Title: Diagnostic Value of Digital Video Oculography in Patients With White Matter Lesions
Brief Title: Diagnostic Value of eVOG
Acronym: DIVEyes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-PP-08
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Radiologically Isolated Syndrome; White Matter Lesions
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- suggestive demyelinating disease (Other): White matter lesions suggestive demyelinating diseases
  Interventions: Procedure: eVOG
- no suggestive demyelinating diseases (Other): White matter lesions not suggestive demyelinating diseases
  Interventions: Procedure: eVOG
- Controls (Other): patients controls
  Interventions: Procedure: eVOG

INTERVENTIONS:
Procedure: eVOG — video digital oculography

SUMMARY:
Eye movement is a complex neurological function controlled by many structures located in the central nervous system. The eyeball is mobile within the orbit and its movements are carried out using 6 muscles innervated by 3 oculomotor nerves allowing to perform reflex or voluntary eye movements in all elementary directions.

So-called internuclear structures allow the two eyeballs to perform combined movements. The attack of these structures during an acute or chronic neurological disease will most often cause oculomotor paralysis in one or more directions of gaze which will be perceived by the patient as double vision.

So-called supranuclear structures make it possible to generate different types of eye movements: saccades, which are extremely rapid eye movements of very short duration, eye pursuit, which is a slow movement whose purpose is to follow a moving visual target and finally, certain neural circuits are intended to stabilize the gaze.

Many neurological diseases can be accompanied by oculomotor abnormalities affecting saccades or ocular pursuit. These include neurodegenerative diseases characterized by diffuse neurological damage.

Involvement of gaze stabilization structures is also frequently found in certain neurological diseases affecting the posterior fossa.

The clinical examination of oculomotricity focuses mainly on the analysis of ocular mobility in the different directions of space by asking the subject to fix an object (for example a pen) or the index of the examiner in moving in different directions in space. During a classic clinical examination, it is then possible to detect anomalies such as oculomotor paralysis or nystagmus, it is however very difficult to assess the speed or the precision of the saccades, as well as the quality of the pursuit ocular.

As a result, the development of techniques to accurately record eye movements has emerged as a need in order to help in the diagnosis of certain visual disorders and certain neurodegenerative diseases.

Video oculography (VOG) is a technique for precisely recording and analyzing the movements of the eyeballs.

The use of VOG in neurology has long been dominated by helping to diagnose certain neurodegenerative diseases and in particular certain atypical Parkinson's syndromes. The value of VOG has also been demonstrated in certain pathologies characterized by atrophy of the brainstem or cerebellum, of hereditary or acquired origin. Some studies have also assessed its contribution to the diagnosis and management of certain dementias and certain psychiatric diseases such as schizophrenia. More recently, the interest of VOG has also emerged in the management of patients with a demyelinating disease of the multiple sclerosis spectrum.

The VOG has a number of limitations to its large-scale use, first of all, it is an examination requiring specific, relatively expensive equipment. On the other hand, the examination requires know-how, both for the passing of the tests but also for the processing and analysis of the data.

The eVOG (mobile VideoOculoGraphy) application has been developed to record oculomotor movements during different paradigms: horizontal saccades, vertical saccades, antisaccades, horizontal pursuit, vertical pursuit thanks to a tablet fixed on a support allowing keep in a stable and fixed position.

The eVOG app was compared to a conventional VOG platform in a first study. The objective was to compare the measurements obtained by the eVOG application to the measurements collected by the standard method in a sample of patients with multiple sclerosis. This study showed that the detection of different anomalies by eVOG is correlated with classic VOG.

In view of these encouraging preliminary results, a prospective study could be set up with the objective of evaluating the value of digital VOG in the diagnostic process in patients referred to a tertiary center for white matter signal abnormalities on MRI.

the hypothesis is that subclinical oculomotor disorders will be found more frequently in the group of patients with MS spectrum disease due to the presence in this pathology of diffuse inflammatory and degenerative damage to brain tissue, unlike the others inflammatory or non-inflammatory pathologies.

ELIGIBILITY:
Patients Inclusion Criteria:

* Patients referred to our tertiary center for a diagnostic workup of white matter hypersignals
* Absence of oculomotor disorders on conventional clinical examination
* Age > 18 years

controls Inclusion criteria:

* The controls can be recruited from the accompanying persons of the patients selected for the study, from the staff of the CHU of Nice or from the entourage of the investigating team;
* Absence of known oculomotor disorders by the control
* Age > 18 years

Exclusion Criteria:

* Presence of a neurological, ophthalmological or general pathology that may interfere with the performance of digital video oculography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
interest of digital VOG at the diagnostic stage in patients referred to a tertiary center for discovery on MRI of white matter lesions. (square wave jerks) | day of inclusion
  The interpretation of the VOG will reveal the presence or absence of the following eye movement abnormalities (EMA):
  - Presence of square wave jerks 0 or 1
interest of digital VOG at the diagnostic stage in patients referred to a tertiary center for discovery on MRI of white matter lesions. (Horizontal saccades abnormalities) | day of inclusion
  The interpretation of the VOG will reveal the presence or absence of the following eye movement abnormalities (EMA):
  - Presence of Horizontal saccades abnormalities 0 or 1
interest of digital VOG at the diagnostic stage in patients referred to a tertiary center for discovery on MRI of white matter lesions. (Vertical saccades abnormalities) | day of inclusion
  The interpretation of the VOG will reveal the presence or absence of the following eye movement abnormalities (EMA):
  - Presence of Vertical saccades abnormalities 0 or 1
interest of digital VOG at the diagnostic stage in patients referred to a tertiary center for discovery on MRI of white matter lesions. (Smooth pursuit abnormality) | day of inclusion
  The interpretation of the VOG will reveal the presence or absence of the following eye movement abnormalities (EMA):
  - Presence of Smooth pursuit abnormality 0 or 1
interest of digital VOG at the diagnostic stage in patients referred to a tertiary center for discovery on MRI of white matter lesions. (Antisaccade abnormality) | day of inclusion
  The interpretation of the VOG will reveal the presence or absence of the following eye movement abnormalities (EMA):
  - Antisaccade abnormality 0 or 1
interest of digital VOG at the diagnostic stage in patients referred to a tertiary center for discovery on MRI of white matter lesions | day of inclusion
  score (0 to 5) of he interpretation of the VOG will reveal the presence or absence of the following eye movement abnormalities (EMA)

SECONDARY OUTCOMES:
Correlations between the presence of EMA and the diffuse damage to brain tissue measured by MRI.(In the subgroup of patients with RIS, CIS or MS, to study) | day of inclusion
  Global and regional volumetric measurements
association between the number or type of EMA at inclusion and the occurrence of a clinical conversion to multiple sclerosis (EDSS) | each year to 2 years
  EDSS score
association between the number or type of EMA at inclusion and the occurrence of a clinical conversion to multiple sclerosis (second line treatment) | at year 1 and year 2
  Evolution towards an active form requiring the use of a second-line treatment (natalizumab, ocrelizumab, fingolimod, cladribine)
association between the number or type of EMA at inclusion and the occurrence of a clinical conversion to multiple sclerosis (secondary progressive form) | at year 1 and year 2
  Evolution towards a secondary progressive form (clinically)
type of EMA between patients and controls | day of inclusion
  type of EMA
number of EMA between patients and controls | day of inclusion
  Number of EMA

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No